CLINICAL TRIAL: NCT01479972
Title: Phase II Open Label, Randomized, Controlled Study to Evaluate Safety and Immunogenicity of VPM1002 in Comparison With BCG in HIV-unexposed, BCG Naive Newborn Infants in South Africa
Brief Title: Study to Evaluate Safety and Immunogenicity of VPM1002 in Comparison With BCG in Newborn Infants in South Africa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Serum Life Science Europe GmbH (Industry)
Collaborators: Children's Infectious Diseases Clinical Research Unit (KID-CRU), South Africa (Unknown); Triclinium Johannesburg, South Africa (Unknown); University of Stellenbosch (Other); HJ-CTC George, South Africa (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VPM1002-ZA-2.12TB; DOH-27-0911-3677 (Other: NHREC (National Health Research Council) South Africa)
Record Dates: First submitted 2011-11-18; First posted 2011-11-28 (Estimated); Last update posted 2013-10-29 (Estimated); Status verified 2013-10

CONDITIONS: Tuberculosis
Keywords: Tuberculosis; Vaccine; Live vaccine; rBCG
MeSH Terms: conditions — Tuberculosis | interventions — VPM1002 recombinant BCG vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VPM1002 (Experimental)
  Interventions: Biological: VPM1002
- BCG (Active Comparator)
  Interventions: Biological: BCG

INTERVENTIONS:
Biological: VPM1002 — Tuberculosis vaccine
  Arms: VPM1002
Biological: BCG — commercially available live vaccine BCG
  Arms: BCG

SUMMARY:
Goal of VPM is the development of a recombinant urease C-deficient listeriolysin expressing BCG vaccine strain (VPM1002) as a safe, well tolerated and efficacious vaccine against tuberculosis (TB) for residents in endemic areas and persons at risk in non-endemic areas. The new vaccine should be at least as potent as the current strain and should be safer than BCG (Kaufmann, 2007a; Grode et al., 2005). The vaccine is formulated as live lyophilised bacteria to be re-suspended before intradermal injection. The preceding clinical trials in 80 volunteers in Germany and 24 volunteers in Bloemfontein, South Africa indicated immunogenicity and safety being sufficient for proceeding with the clinical development in newborn infants. Hence, the current study is commenced at Stellenbosch University, South Africa. This is the first investigation of VPM1002 in newborn infants.

ELIGIBILITY:
Inclusion Criteria:

Maternal:

1. The infant's mother must be aged 18 years or older at the time of screening.
2. The infant's mother must be able and willing to comply with the study protocol, available and willing to allow her child to complete all the study assessments and must have signed an Informed Consent form that has been approved by all relevant Ethics Committee/s.
3. The infant's mother must not have any symptoms or signs of either active TB or latent tuberculosis infection as indicated by:

   * History of cough for more than two weeks, fever, weight loss, breathlessness, chest pain, blood in sputum, night sweats and loss of appetite, and/or
   * Mantoux Tuberculin PPD skin test greater than or equal to 10 mm
4. The infant's mother should not be planning to relocate from the research site area and should be reachable by phone during the whole study period i.e. for the 6 month on-study period as well as the 30 month structured medical surveillance period.
5. The infant's mother must test negative for HIV-1 (ELISA 4th generation) within the period from 2 weeks prior to the infant's birth to vaccination of the infant with the investigational product.
6. The infant's mother must test negative for Hepatitis B and Syphilis serology at screening.
7. The infant's mother should have no history or evidence of Diabetes Mellitus.
8. No participation of the infant's mother in a clinical trial within 3 months prior to the birth of the participating infant. In addition, if breast-feeding, no participation in another clinical trial during the 6 months of the current study.
9. The infant's mother must have no known history of immunodeficiency.

Infant:

1. Healthy full-term male or female newborn infants aged 0 to 8 days.
2. Infants must have a birth weight of 3000 - 4000 g and an Apgar score of > 9 at 5 minutes.
3. No eczema or other significant skin lesion or infection at the intended injection site.
4. No routine BCG vaccination administered (as per vaccination record)
5. Infants must have received Oral Polio Vaccine as part of the routine South African Expanded Programme on Immunisation (EPI) Childhood Immunisation schedule, and must adhere to the subsequent EPI schedule for the entire study period, except for the BCG vaccination at birth.
6. No participation of the infant in another clinical trial before study vaccination and during the 6 months of the current study.

Exclusion Criteria:

Maternal:

1. Known presence of any person in the household of the mother and newborn infant, or any visitor to the household with reported active tuberculosis disease.
2. Treatment of the mother with blood products in the 6 months prior to or during the birth of the participating infant.
3. Positive test for HIV-1 either during the current pregnancy or at screening.
4. Positive screening test for Hepatitis B or Syphilis.
5. History or evidence of Diabetes Mellitus.
6. Presence of any symptoms or signs of either active TB or latent tuberculosis infection as indicated by:

   * History of cough for more than two weeks, fever, weight loss, breathlessness, chest pain, blood in sputum, night sweats and loss of appetite, and/or
   * Mantoux Tuberculin PPD skin test greater than or equal to 10 mm (read 48-72hrs post-test)
7. Presence of signs or symptoms of any reported acute infectious disease at the time of screening.
8. Any reported or suspected substance abuse.

Infant:

1. History or evidence of any systemic disease on physical examination or any acute, chronic or intercurrent illness that, in the opinion of the investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.

   Note: Neonatal jaundice which is not considered by the investigator to be clinically significant will not represent exclusion.
2. Vaccination with routine BCG before study vaccination.
3. Fever within the period post birth and prior to dosing. For the purposes of this protocol, fever in the infant will be defined as an axillary body temperature > 38.0°C measured with a digital thermometer on at least 2 occasions not less than 6 hours apart.
4. Hypothermia within the period post birth and prior to dosing. For the purposes of this protocol, hypothermia in the infant will be defined as an axillary body temperature < 36.0°C measured with a digital thermometer on at least 2 occasions not less than 6 hours apart.
5. Clinically suspected neonatal sepsis.
6. Any malignant condition.
7. Any severe congenital malformation.
8. Concomitant treatment with medication that may significantly affect immune function (e.g. systemic corticoids, immunosuppressive drugs) before study vaccination. Antibiotics given before study vaccination would further constitute exclusion.
9. Treatment of the infant with blood products.
10. Any clinically significant laboratory abnormalities on screening blood samples or urinalysis.

Max Age: 8 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Safety | Six months
  Safety and tolerability as assessed by monitoring of adverse events (incidence, time profile, other profiles, and including local or regional reactions at the vaccination site), physical examination, vital signs, standard laboratory safety parameters, including haematology, clinical chemistry and urinalysis.

SECONDARY OUTCOMES:
Immunogenicity | baseline, day 14, week 6, 12, 18, month 6
  IFN-gamma-WB-ELISA: concentration of IFN-gamma per ml supernatant after stimulation. ICS (FACS): number of CD4+ T-lymphocytes ("single-positive-cells", "double-positive-cells", "triple-positive-cells", "multi-positive-cells (positive for at least two of IFN-gamma, TNF-alpha or IL-2) after 16 hours stimulation; per total number of lymphocytes. ICS (FACS): number of CD8+ T-lymphocytes("single-positive-cells", "double-positive-cells", "triple-positive-cells", "multi-positive-cells (positive for at least two of IFN-gamma, TNF-alpha or IL-2) after 16 hours stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cotton, MD, Professor, Principal Investigator — Children's Infectious Diseases Clinical Research Unit (KID-CRU), Tygerberg, South Africa
Locations (1):
- Children's Infectious Diseases Clinical Research Unit, Tygerberg Hospital, Cape Town, South Africa

REFERENCES:
- [Derived] Loxton AG, Knaul JK, Grode L, Gutschmidt A, Meller C, Eisele B, Johnstone H, van der Spuy G, Maertzdorf J, Kaufmann SHE, Hesseling AC, Walzl G, Cotton MF. Safety and Immunogenicity of the Recombinant Mycobacterium bovis BCG Vaccine VPM1002 in HIV-Unexposed Newborn Infants in South Africa. Clin Vaccine Immunol. 2017 Feb 6;24(2):e00439-16. doi: 10.1128/CVI.00439-16. Print 2017 Feb. PMID 27974398